CLINICAL TRIAL: NCT07360769
Title: Low Dialysate Flow: Its Effect on Hemodialysis Adequacy, Dialysis Recovery Time and Patient Reported Outcome Measures.
Brief Title: Optimizing Hemodialysis: How Low Dialysate Flow Alters Adequacy and Patient Recovery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0108861
Record Dates: First submitted 2025-12-15; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-03

CONDITIONS: End Stage Kidney Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESKD patients (Active Comparator)
  Interventions: Other: lower dialysate flow rate ( 300ml/min). then testing its effect on hemodialysis adequacy

INTERVENTIONS:
Other: lower dialysate flow rate ( 300ml/min). then testing its effect on hemodialysis adequacy — The aim of this study is to check whether change of dialysate flow from 500ml/min to 300ml/min has a significant impact on dialysis adequacy , dialysis recovery time and patient reported outcome measures in maintenance hemodialysis patients.

SUMMARY:
The goal of this clinical trial is to detect if lower dialysate flow rate can affect hemodialysis adequacy , dialysis recovery time and patients quality of life.

The main questions it aims to answer are:

does low dialysate flow affect hemodialysis adequacy? does green dialysis achievable without affecting hemodialysis adequacy? Researchers will compare hemodialysis session of high dialysate flow to that with low dialysate flow.

Participants will:

underwent hemodialysis for a week with low dialysate flow and another week with high dialysate flow.

ELIGIBILITY:
Inclusion Criteria:

* ESKD patients more than or equal 18 years old, on maintenance HD thrice weekly for more than three months and each session lasts for 4 hours.
* All patients will receive HD via an arterio-venous fistula.
* All patients will receive HD via the same type of HD machine and the blood pump will be set at 300ml/min.
* All patients will receive the same type of HD membranes and every effort will be made to achieve the dry weight of the patients.

Exclusion Criteria :

* Critically ill and hospitalized ESKD patients.
* Mentally disabled patients.
* Patients with terminal malignancy or receiving chemotherapy.
* Patients receiving immune suppression treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
The change of dialysate flow rate, for three successive conventional hemodialysis sessions, from 500ml/min to 300ml/min and its impact on hemodialysis adequacy that is assessed by urea reduction ratio (URR). | Two weeks
The change of dialysate flow rate, for three successive conventional hemodialysis sessions, from 500ml/min to 300ml/min and its impact on hemodialysis adequacy that is assessed by and single-pool Kt/V (spKt/V) using the Daugirdas formula. | Two weeks

SECONDARY OUTCOMES:
The effect of lowering dialysate flow rate from 500ml/min (milli per minute) to 300ml/min on dialysis recovery time (DRT) in minutes. Longer duration indicates lower dialysis adequacy. | two weeks
The patients reported outcome measures that is assessed by palliative care Outcome Scale - Symptoms Renal (POS S renal). Each symptom takes a score from zero to four (0-4), high score indicates less efficient dialysis. | Tow weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided